CLINICAL TRIAL: NCT01840033
Title: A Monocenter Prospective Study to Evaluate the Efficacy of Peripherally Inserted Central Catheter to Tunnelled Central Catheter With Cuff in Home Parenteral Nutrition for Long-term Used: the PICCnut Study.
Brief Title: A Monocenter Prospective Study to Evaluate the Efficacy of Peripherally Inserted Central Catheter to Tunnelled Central Catheter With Cuff in Home Parenteral Nutrition for Long-term Used.
Acronym: PICCNUT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of selection of inclusion
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-PP-02
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Chronic Intestinal Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group B (Active Comparator): After consent, patients will be randomised to PICC Line (group A) or tunnelled nutritional central catheter with cuff (group B). Duration of inclusion will be 24 months. After randomisation, patients will have catheter inserted by a competent radiologist following an echography. Radiologist will have to answer a questionnaire and doctors will note any catheter-related complications.
  Interventions: Device: Tunnelled nutritional central catheter
- Group A (Experimental): PICC Line (group A) : patients will have catheter inserted by a competent radiologist following an echography. Radiologist will have to answer a questionnaire and doctors will note any catheter-related complications.
  Interventions: Device: group Piccnut

INTERVENTIONS:
Device: group Piccnut — Vessels echography will be systematically repeated at 3 months and 12 months for thrombosis research. Follow-up visit will be held at 1,3,6,9 and 12 months. At every step, major and minor complications will be noted by the investigators.
  Arms: Group A
Device: Tunnelled nutritional central catheter — After consent, patients will be randomised to PICC Line (group A) or tunnelled nutritional central catheter with cuff (group B). Duration of inclusion will be 24 months. After randomisation, patients will have catheter inserted by a competent radiologist following an echography. Radiologist will have to answer a questionnaire and doctors will note any catheter-related complications. After that, vessels echography will be systematically repeated at 3 months and 12 months for thrombosis research. Follow-up visit will be held at 1,3,6,9 and 12 months. At every step, major and minor complications will be noted by the investigators.
  Arms: Group B

SUMMARY:
Home parenteral nutrition (HPN) is the reference treatment for anatomic or fonctionnal chronic intestinal failure. Nutritionnal catheter must follow two rules: low infection rate and be able to preserve the permeability of the central vein. Today, in europeen guidelines, two types of central devices are recommended: tunnelled central catheter with cuff and implanted ports. However, their insertion is not without risk. Since many years, we have seen a new generation of catheter - peripherally inserted central catheter (PICC line)- which have many advantage over other central catheter. ESPEN guidelines accept the use of PICC line in short and moderate-term for HPN, but no prospective study have look for long-term used in HPN.

The objective of our study is to evaluate in a prospective randomised monocenter study the no-inferiority of PICC line to tunnelled central catheter with cuff for serious catheter related-complications such as infection and thrombophlebitis for patient on HPN over 1 month of duration. The secondary objectives are to: evaluate the number of patients with at least one serious complications related in 1000 days of used, the rate of minors and majors complications, number of catheter inserted, the satisfaction of patients and doctors.

The study is held in CHU Nice and will be proposed to hospitalized patients who will need HPN. After consent, patients will be randomized to receive PICC Line (group A) of nutritional central catheter with cuff (group B). Echography of vessels will be held at the beginning, 3 months and 12 months. Follow-up will be conduct at regular interval (month 0-1-3-6-9-12). The duration of follow-up will be of 12 months and the global duration of the study will be 36 months. One major complication will conduct to withdrawal of the study. There will be 55 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years-old
* Patients managed by CHU Nice for home parenteral nutrition
* Expected to have over 1 month of parenteral nutrition
* Signed consent
* Affiliation to Securite Social

Exclusion criteria

* Patient with nutritional catheter before inclusion
* Pregnancy or breastfeeding
* Evolutive pathology with life expectancy < 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
major complications | 12 months
  Statically significative difference between rate of incidence of major complications (infection and/or thrombosis related to catheter) during the 12 months follow-up.

SECONDARY OUTCOMES:
Delay | 12 months
  Delay in days between insertion and first major complications
Questionnaire | 12 months
  Questionnaire to evaluate catheter insertion by radiologist (satisfaction and complications).
  Satisfaction questionnaire to patients at every visit

CONTACTS AND LOCATIONS:
Overall Officials: HEBUTERNE Xavier, PhD, Principal Investigator — CHU de Nice, Hôpital Archet, Pôle Digestif, 151 route de saint-antoine de ginestière 06200 Nice
Locations (1):
- CHU de Nice, Nice, Alpes-Maritimes, France